CLINICAL TRIAL: NCT05001529
Title: Flow Cytometry Analysis of Eosinophils Activity and Membrane Receptors Expression in Severe Asthma Patients: Basal Characterization and Evaluation of Changes Induces by Biological Drugs.
Brief Title: Flow Cytometry Analysis of Eosinophils in Severe Asthma Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scarlata, Simone, M.D. (Other)
Collaborators: IRCCS San Raffaele (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EoAG
Record Dates: First submitted 2021-04-23; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Severe Asthma
Keywords: severe asthma; eosinophils phenotype; anti-IL5R antibody
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Subject with severe asthma, treated with anti IL5R antibodies
  Interventions: Biological: anti IL5 receptor antibodies
- Group B (No Intervention): Subject with severe asthma, treated with conventional therapy

INTERVENTIONS:
Biological: anti IL5 receptor antibodies — Subjects with severe uncontrolled asthma will be assigned to treatment with Omalizumab (anti Ig E antibodies) or Mepolizumab (anti IL-5 antibodies) according to medical advice and standardized protocols for asthma treatment.
  Arms: Group A

SUMMARY:
Asthma is a heterogeneous disease, characterized by reversible airflow obstruction, airway hyperresponsiveness, and airway inflammation, in which 40% of patients exhibit eosinophil-driven pathobiology.The main treatment of asthma is the use of corticosteroid, whose use induces a reduction in eosinophils that is considered a strong predictor of response to treatment. Corticosteroids have remained the mainstay treatment of asthma and reduction in eosinophils has remained the unequivocal predictor of steroid response. The prevalence of asthma, which is expected to increase, it is about 300 million people worldwide. About 5-10% of asthma patients have severe disease, which is defined as asthma that requires high-dose inhaled corticosteroids (ICSs) plus a second controller to prevent it from becoming "uncontrolled" or which remains "uncontrolled" despite this therapy. Patients with severe disease have worse quality of life, and disproportionately high morbidity, mortality, and use of health care resources when compared with their peers with well-controlled disease.The pathophysiology of asthma is complex and heterogeneous between patients, as the disease itself; however, on the basis of immune system involvement, it is possible to define 2 subtypes - or endotypes- of asthma. These endotypes are named T2 (for type 2 cells) high or low, and are defined by the levels of expression of the T2 cytokines, IL-4, IL-5, and IL-13 produced by T helper 2 lymphocytes, and innate lymphoid cell-2.T2 high endotype patients display an increase in the number of blood and sputum eosinophils, and have a better response to the current available biological therapies , such as the administration of mepolizumab (anti IL-5 antibody). Eosinophilic asthma is associated to a more severe clinical phenotype,but patients with a T2 endotype respond better to biological therapies. The hypothesis of the present proposal is that the activation status of these cells, analyzed by the expression of activation markers, can be used to define a new, different, endotype, in which eosinophils, although quantitatively low or normal, are qualitatively more active and aggressive, and could therefore act as an indicator of the progression toward a T2 high endotype.Moreover, the investigators will verify whether a different expression of these molecules on eosinophil's surface might be associated with different clinical response to biologic medications.

DETAILED DESCRIPTION:
Subject satisfying eligibility criteria will be asked to participate the study; all will receive a detailed explanation of the nature of the study, of the aims and objectives. After having signed informed consent, patients will be divided into two groups, based on their clinical status: controlled asthma group (group A) and severe asthma group (group B). Visits will be planned at recruitment, after a run-in period (3-months), meant to optimize first and second lines medical treatment and confirm diagnosis of severe asthma. After the run-in period, patients will be re-evaluated and appropriate medical therapy will be tailored (T0). To group B, therapy with Mepolizumab or Omalizumab will be given, according to standard guidelines. At T0 a blood sample will be collected (3ml) to evaluate eosinophils phenotype by flow cytometry (see below). After 6 months (T1/2) and12 months (T1) patients will be visited again and a blood sample will be taken for flow cytometry analysis.All samples will be properly stored and shipped for analysis, according to best of practice and state of art criteria, within 6 hours from sample's collection. Data will be collected and stored according to the GDPR (General Data Protection Regulation, EU 2016/679). Biological material collected will be used only for the indicated assay and excess material will be discharged.

* Baseline evaluation (T'0) In case of acceptance, and after signing an informed consent, participants will be asked to collect a complete medical history, including allergies and Asthma related comorbidities; a comprehensive physical examination and respiratory function tests consisting of: flow-volume spirometry plus residual volume and DLCO determination. In case of a first diagnosis of asthma a bronchodilator response or a methacholine challenge tests will be obtained. In case of a preexistent diagnosis of asthma, previous examination confirming and proving the diagnosis will be collected.
* Evaluation Tool The following data will be collected at T'0, T'1/2 (six months) and T'1 (twelve months): Clinical assessment: ACT, on demand or rescue therapy, acute exacerbations, medical visits, working absences, hospital admissions. Functional assessment: Flow volume curve, Residual volume, Ig E and eosinophils' count, FeNO, 6 minutes walk test.
* Flow cytometry The investigators will evaluate, by multicolor flow cytometry, the expression of molecules on eosinophils'membrane, using a whole-blood staining protocol, so that blood samples will be minimally manipulated, thus reducing the possibility of artifacts. Briefly, peripheral blood samples will be processed within 6 hours from withdrawal. Samples will be stored at room temperature until processing. Blood samples will be stained, using fluorochrome conjugates antibodies directed towards eosinophils'surface molecules. In particular, the investigators will use antibodies against CD45, CD66, CD15, CD16 and Siglec-8, which will be used to identify eosinophils between other leukocytes; CD63, CD294 (CRTH2, prostaglandin D2 receptor), CD125 (IL-5 receptor), CD193 (receptor for several chemokines, as for example RANTES, Eotaxin, MCP-3, MIP1α), and HLA-DR: these molecules are upregulated with eosinophils activation, so they can have an altered expression in severe asthma patients. After 30 minutes incubation at 4°C, FACS lysing solution (BD Bioscience) will be used to remove erythrocytes, according to manufacturer's instruction. Samples will be resuspended in phosphate buffered saline (PBS) and acquired on a LSRFortessa X-20 (BD Bioscience) flow cytometer, equipped with four lasers.

ELIGIBILITY:
Inclusion Criteria:

* proved diagnosis of severe, refractory eosinophilic asthma, according to GINA recommendations and International ERS/ATS guidelines;
* agreeing to participate this study and signing an informed consent.

Exclusion Criteria:

* current smoking habit (both tobacco and e-cigarettes),
* concomitant diseases requiring chronic administration of immunosuppressors, biologic medications or systemic corticosteroids for any disease other than asthma
* History of previous or concomitant acute or chronic disease known to directly or indirectly affect eosinophil count, both in a quantitative and qualitative manner (eosinophilic lung and gastrointestinal diseases, systemic vasculitis, allergic bronchopulmonary aspergillosis, parasitic infections, etc)
* COPD/Asthma overlap.
* Inability or denial to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Measurement by flow cytometry of differences in the percentages of eosinophils expressing activation-related molecules | 12 months
  The presence of activated eosinophils will be evaluated by flow cytometry analysis of the expression of CD193, CD63, CD294, CD125, and HLA-DR on eosinophils membrane.
  Results will be expressed in term of percentage (%) of eosinophils expressing the molecules;
Measurement by flow cytometry of the expression levels of activation markers on eosinophils membrane | 12 months
  Activation-associated membrane markers (CD193, CD63, CD294, CD125, and HLA-DR) on eosinophils membrane will be evaluated by flow cytometry and results will be expressed in term of Mean Fluorescence intensity (MFI) of the molecules. MFI is a measure of the amount of the molecule expressed on eosinophils membrane: the higher the MFI, the higher the density of molecules on cellular membrane.
  The values will be expressed as arbitrary units (AU), defined by the instrument, comparing the samples with a negative (unstained) control.

SECONDARY OUTCOMES:
Correlation between activated eosinophils phenotype and disease progression | 12 months
  Statistical analysis will be used to define the possible correlation between expression of activation markers on eosinophils (as described in primary outcomes 1 and 2) and the clinical status of the patients, evaluated by Flow volume curve, Residual volume, Ig E and eosinophils' count, 6 minutes walking test.
Change in the percentage of activated eosinophils in the group of patients receiving the biological treatment. | 12 months
  Flow cytometry analysis of eosinophils will be performed before and after one year of treatments with antibodies against IL-5 or IL-5R. Percentages of activated eosinophils will be measured as described in Primary outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Campus Bio Medico University and Teaching Hospital, Roma, Italy